CLINICAL TRIAL: NCT03613142
Title: Comparison Between Double Tract Anastomosis and Esophagogastrostomy After Radical Proximal Gastrectomy: A Prospective, Randomized, Controlled Study
Brief Title: Comparison Between Double Tract Anastomosis and Esophagogastrostomy After Radical Proximal Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Biao Fan, MD, Clinical Professor, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: DTvsEG
Record Dates: First submitted 2018-07-23; First posted 2018-08-02 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer
Keywords: Double tract; Esophagogastrostomy; Gastric cancer; GastroEsophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double tract anatomosis (Experimental): After the proximal gastrectomy, the purse-string suture is tied at the esophagus stump, and the anvil head is inserted into the esophagus stump using an anvil clamp. A Roux-en-Y esophagojejunostomy (E-stomy) is performed by intracorporeal anastomosis with a circular stapler, and the jejunal stump is closed with a linear stapler. Next, side-to-side gastrojejunostomy (G-stomy), 15 cm below the E-stomy, is performed using 2 linear staplers. Finally, end-to-side jejunojejunostomy (J-stomy), 20 cm below the G-stomy, is performed by 2 linear staplers.
  Interventions: Procedure: Double tract anatomosis
- Esophagogastrostomy (Active Comparator): After the proximal gastrectomy, the purse-string suture is tied at the esophagus stump, and the anvil head is inserted into the esophagus stump using an anvil clamp. Next, end-to-end or side to end esophagogastrostomy is performed with a circular stapler.
  Interventions: Procedure: Esophagogastrostomy

INTERVENTIONS:
Procedure: Double tract anatomosis — After the proximal gastrectomy, the purse-string suture is tied at the esophagus stump, and the anvil head is inserted into the esophagus stump using an anvil clamp. A Roux-en-Y esophagojejunostomy (E-stomy) is performed by intracorporeal anastomosis with a circular stapler, and the jejunal stump is closed with a linear stapler. Next, side-to-side gastrojejunostomy (G-stomy), 15 cm below the E-stomy, is performed using 2 linear staplers. Finally, end-to-side jejunojejunostomy (J-stomy), 20 cm below the G-stomy, is performed by 2 linear staplers.
  Arms: Double tract anatomosis
Procedure: Esophagogastrostomy — After the proximal gastrectomy, the purse-string suture is tied at the esophagus stump, and the anvil head is inserted into the esophagus stump using an anvil clamp. Next, end-to-end or side to end esophagogastrostomy is performed with a circular stapler.
  Arms: Esophagogastrostomy

SUMMARY:
The patients with upper gastric cancer (cT1N0M0) or gastroesophageal adenocarcinoma (diameter less than 4 cm) will be enrolled into this study. Each of these patients will undergo radical proximal gastrectomy and be randomly allocated into one of the two groups, double tract anastomosis group or esophagogastrostomy group. The following data will be collected to compare the difference between the two reconstruction methods: the rate of reflux esophagitis, postoperative quality of life, economic expenditure, the safety of operation, postoperative recovery, postoperative nutrition status and oncological effect. Through the comprehensive analysis, the result of this study will elucidate the best of the reconstruction method after proximal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as gastric or esophagogastric adenocarcinoma
2. Age ranges from 18 to 80
3. Karnofsky assessment no less than 70
4. Completion of abdominal CT scan and ultrasound endoscopy
5. Upper gastric cancer (cT1N0M0) or esophagogastric adenocarcinoma (diameter no more than 4 cm)
6. radical proximal gastrectomy
7. Normal blood routine examination and biochemical test

Exclusion Criteria:

1. Patients need to undergo total gastrectomy or distal gastrectomy
2. Female patients with pregnancy
3. Not suitable for operation
4. Patients have already joined other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of reflux esophagitis after operation | 12 months
  The rate of reflux esophagitis after operation will be assessed by gastrointestinal endoscopy with Los Angeles (LA) classification. the degree of reflux esophagitis will be classified as N, A, B, C or D level, and latter levels represent a more severe reflux esophagitis.

SECONDARY OUTCOMES:
postoperative quality of life | 12months
  Assessed by European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) - C30 questionnaire, the total score ranges from 30 to 126, and higher values represent a worse outcome.
postoperative quality of life | 12months
  Assessed by European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) - STO22 questionnaire, the total score ranges from 22 to 88, and higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Ji, M.D., Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: No